CLINICAL TRIAL: NCT01197573
Title: Enhancing DCD Utilization With Thrombolytic Therapy
Brief Title: Enhancing Donated After Cardiac Death (DCD) Utilization With Thrombolytic Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Bijan Eghtesad, MD, HPBT Staff Surgeon, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CCIRB: 10-365; R38OT15491 (Other Grant/Funding Number: HRSA)
Record Dates: First submitted 2010-09-08; First posted 2010-09-09 (Estimated); Results first posted 2018-08-28 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-07

CONDITIONS: Liver Transplantation; Kidney Transplantation
MeSH Terms: interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Standard DCD liver transplant (Active Comparator): Standard method of liver transplant utilizing a DCD organ
  Interventions: Other: No TPA Treatment
- rTPA Treatment Liver Transplant (Active Comparator): Ex-vivo treatment of liver donated after cardiac death (DCD) with rTPA
  Interventions: Drug: rTPA Treatment
- Standard DCD kidney transplant (Active Comparator): Standard method of kidney transplant utilizing a DCD organ
  Interventions: Other: No TPA Treatment
- rTPA Treatment Kidney Transplant (Active Comparator): Ex-vivo treatment of kidney donated after cardiac death (DCD) with rTPA
  Interventions: Drug: rTPA Treatment

INTERVENTIONS:
Drug: rTPA Treatment — Ex-vivo treatment of DCD liver or kidney with rTPA (recombinant tissue plasminogen activator)prior to implantation
  Other Names: Alteplase
  Arms: rTPA Treatment Kidney Transplant; rTPA Treatment Liver Transplant
Other: No TPA Treatment — Standard of Care
  Arms: Standard DCD kidney transplant; Standard DCD liver transplant

SUMMARY:
We hypothesize that delayed graft function and ITBS events may be related to small blood clots (microthrombi) that collect in the kidneys and liver after cardiac death. Treatment of the DCD organs with a thrombolytic agent prior to implantation may reduce post-transplant morbidity and mortality, and may ultimately result in a greater number of transplantable livers and kidneys.

DETAILED DESCRIPTION:
The waiting list for kidney and liver transplantation continues to increase in the United States, and therefore the need grows for additional donor organs. Utilization of organs donated after cardiac death (DCD) could be one way to increase organ availability, however there are risks associated with poorer clinical outcomes, including delayed graft function and in livers specifically, ischemic-type biliary strictures (ITBS). We hypothesize that delayed graft function and ITBS events may be related to small blood clots (microthrombi) that collect in the kidneys and liver after cardiac death. Treatment of the DCD organs with a thrombolytic agent prior to implantation may reduce post-transplant morbidity and mortality, and may ultimately result in a greater number of transplantable livers and kidneys.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older
* Subjects willing/able to provide written consent
* Subjects willing/able to comply with study requirements
* Subjects who will receive a solitary organ transplant

Exclusion Criteria:

* Subjects requiring multi-organ transplants
* Women who are pregnant
* Subjects with current severe systemic infection
* Subjects with an active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2010-04; Primary Completion 2015-10 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bijan Eghtesad, MD, Principal Investigator — The Cleveland Clinic
Locations (2):
- United States (2):
  - University Hospitals / Case medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: DCD donors from 2010 to 2013.
Groups:
- rTPA Treatment - Liver: Ex-vivo treatment of liver donated after cardiac death (DCD)with rTPA
  rTPA Treatment: Ex-vivo treatment of DCD liver with rTPA (recombinant tissue plasminogen activator)prior to implantation
- rTPA Treatment - Kidney: Ex-vivo treatment of kidney donated after cardiac death (DCD)with rTPA
  rTPA Treatment: Ex-vivo treatment of DCD kidney with rTPA (recombinant tissue plasminogen activator)prior to implantation
Period: Overall Study
Arm/Group | Standard DCD Liver Transplant | rTPA Treatment - Liver | Standard DCD Kidney Transplant | rTPA Treatment - Kidney
Started | 33 | 46 | 12 | 12
Completed | 33 | 46 | 12 | 12
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard DCD Liver Transplant | rTPA Treatment - Liver | rTPA Treatment - Kidney | Standard DCD Kidney Transplant | Total
Number analyzed (Participants) | 33 | 46 | 12 | 12 | 103
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 33 | 46 | 11 | 11 | 101
  >=65 years | 0 | 0 | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 15 | 4 | 2 | 40
  Male | 14 | 31 | 8 | 10 | 63
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 8 | 5 | 18
  White | 30 | 43 | 4 | 7 | 84
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 33 | 46 | 12 | 12 | 103

OUTCOME MEASURES:

1. Primary Outcome: Delayed Kidney Graft Function
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | rTPA Treatment - Kidney | Standard DCD Kidney Transplant
Number analyzed (Participants) | 12 | 12
Participants | 5 | 7

2. Primary Outcome: Number of Participants With Primary Liver Graft Nonfunction
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Groups:
- rTPA Treatment: Ex-vivo treatment of liver donated after cardiac death (DCD)with rTPA
  rTPA Treatment: Ex-vivo treatment of DCD liver with rTPA (recombinant tissue plasminogen activator)prior to implantation
Arm/Group | Standard DCD Liver Transplant | rTPA Treatment
Number analyzed (Participants) | 33 | 46
Participants | 2 | 1

3. Secondary Outcome: Number of Participants With Liver Ischemic-Type Biliary Strictures
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Standard DCD Liver Transplant | rTPA Treatment
Number analyzed (Participants) | 33 | 46
Participants | 0 | 3

ADVERSE EVENTS:
Time Frame: One Year
Groups:
- Standard DCD Kidneytransplant: Standard method of kidney transplant utilizing a DCD organ
Arm/Group | Standard DCD Liver Transplant | rTPA Treatment - Liver | rTPA Treatment - Kidney | Standard DCD Kidneytransplant
All-Cause Mortality (participants affected / at risk) | 6/33 | 12/46 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 3/33 | 2/46 | 2/12 | 2/12
Other Adverse Events (participants affected / at risk) | 12/33 | 8/46 | 5/12 | 7/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard DCD Liver Transplant (N=33) | rTPA Treatment - Liver (N=46) | rTPA Treatment - Kidney (N=12) | Standard DCD Kidneytransplant (N=12)
Primary non -function (Surgical and medical procedures) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Necrosis (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Necrotic Right Colon
Bleeding (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary Leak (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard DCD Liver Transplant (N=33) | rTPA Treatment - Liver (N=46) | rTPA Treatment - Kidney (N=12) | Standard DCD Kidneytransplant (N=12)
Delayed Graft Function (Surgical and medical procedures) | 12 (12) | 8 (8) | 5 (5) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes